CLINICAL TRIAL: NCT02438358
Title: Feasibility of the LUM Imaging System for Intraoperative Detection of Residual Cancer in the Tumor Bed of Female Subjects With Breast Cancer
Brief Title: Feasibility Study of Intraoperative Imaging in Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lumicell, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Massachusetts General Hospital (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LUM-015/2.6-001; 1R21CA173762 (NIH)
Record Dates: First submitted 2015-04-17; First posted 2015-05-08 (Estimated); Results first posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- LUM Imaging System (Experimental): No dose or a single dose of LUM015 (0.5 mg/kg or 1.0 mg/kg) will be administered by intravenous injection between 2 to 6 hours prior to surgery. The dose administered in Phase B will be determined based on results of Phase A. All subjects will have intraoperative imaging using the LUM 2.6 Imaging Device.
  Interventions: Drug: LUM015; Device: LUM 2.6 Imaging Device

INTERVENTIONS:
Drug: LUM015
Device: LUM 2.6 Imaging Device

SUMMARY:
For most breast cancer patients, surgery is the primary treatment. When patients undergo a lumpectomy, it is difficult for the surgeon to determine the extent of the tumor which results in incomplete tumor removal as determined by a positive margin assessment several days after the initial surgery is completed. Most patients with positive margins will undergo a second or even a third surgery to complete the tumor removal. The investigators hypothesize that the LUM Imaging System can reduce the rates of positive margins and, thus, the rates of second surgeries by identifying microscopic residual cancer in the tumor bed.

This is a non-randomized, open label study to evaluate the safety and efficacy of an intraoperative imaging system, the LUM Imaging System (LUM015 in conjunction with LUM 2.6 Imaging Device), in identifying residual cancer in the tumor bed of female breast cancer subjects. The study is composed of a Feasibility Trial divided into two phases: Phase A (15 total subjects) and Phase B (up to 50 total subjects). During Phase A, 15 subjects will be evaluated to collect additional patient safety data, select the dose of LUM015 for Phase B and evaluate the device function. During Phase B, subjects will be injected with LUM015 at the dose determined during Phase A to preliminarily assess the performance of the detection algorithm against pathology margin assessment. In Phase B, the surgeon will perform standard of care surgery and then use the LUM Imaging System to guide the removal of additional cavity shavings as indicated by the LUM Imaging System.

DETAILED DESCRIPTION:
The LUM Imaging System consists of the cancer imaging agent LUM015 and a hand-held fluorescence-based imager that collects the emission of activated LUM015 in and around tumor. The LUM Imaging System is designed to detect microscopic residual cancer cells in real-time within the tumor bed. In this study, we will evaluate the performance of the LUM Imaging System in detecting residual cancer and guiding its removal during lumpectomies.

In Phase A, all patients will receive standard of care surgery followed by intraoperative imaging of the tumor bed and resected tissue with the LUM 2.6 Imaging Device. In Phase A, no clinical decisions are made based on the imaging results. Standard of care margin assessment will be performed and compared against the imaging results with the LUM Imaging System.

Subjects in Phase B will receive standard of care surgery followed by intraoperative imaging of the tumor bed with the LUM Imaging System. In Phase B, the surgeon will remove an additional shaved margin specimen if indicated by the LUM Imaging System. Final margin assessment will be performed on the very last shaved margin specimen removed.

All participating subjects will be observed to collect safety data from the time of injection of LUM015 to the time the clinical team decides no additional surgery is needed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed primary breast cancer.
* Female, age of 18 years or older.
* Scheduled for a lumpectomy of a breast tumor.
* Able and willing to follow study procedures and instructions.
* Subjects must have received and signed an informed consent form.
* Subjects must be otherwise healthy except for the diagnosis of cancer, as per the exclusion criteria listed below.
* Subjects must have normal organ and marrow function as defined below:

  * Leukocytes > 3,000/mcL
  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
  * Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) starting the day entering the study, and for 60 days after injection of the imaging agent.
* Subjects with ECOG performance status of 0 or 1.

Exclusion Criteria:

* Subjects with a known current condition of substance addiction.
* Subjects who have taken an investigational drug within 30 days of enrollment.
* Subjects with prolonged QT interval.
* Subjects who will have administration of methylene blue or any blue dye used for sentinel node mapping procedures.
* Subjects who have not recovered from adverse events due to pharmaceutical or diagnostic agents administered more than 4 weeks earlier.
* Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 150 mm Hg, or diastolic blood pressure > 95 mm Hg; those subjects with known HTN should be stable within these ranges while under pharmaceutical therapy
* Subjects with insulin dependent diabetes mellitus.
* History of anaphylactic reaction attributed to any contrast agent or drugs containing polyethylene glycol (PEG).
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded. Breastfeeding should be discontinued if the mother is treated with LUM015.
* Subjects who are sexually active and not willing/able to use medically acceptable forms of contraception upon entering the study.
* HIV-positive individuals on combination antiretroviral therapy.
* Any subject for whom the investigator feels participation is not in the best interest of the subject.
* Subjects undergoing a second surgery because they had positive margins in a previous surgery.
* Subjects with prior breast surgeries, mastectomies, breast reconstructions or implants. (Note: subjects who have had prior breast biopsies are not excluded)
* Subjects with prior reduction mammoplasties or breast reductions performed less than 2 years prior to enrollment to this study.
* Subjects previously treated with systemic therapies to treat cancer, such as neo-adjuvant chemotherapy or hormonal therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Smith, M.D., Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase A enrolled 15 women undergoing lumpectomy for primary breast cancers assigned sequentially to one of the 3 different dose arms (no dose of LUM015, 0.5mg/kg of LUM015, and 1.0mg/kg of LUM015).
  Phase B patients enrolled until 10 patients had positive margins in their standard of care cavity shave or a maximum of 50 patients was reached, whichever happened first.
Groups:
- Phase A: No Dose: 5 participants were not injected with LUM015. All subjects will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase A: LUM015 0.5 mg/kg: 5 participants received a single dose of LUM015 0.5 mg/kg administered by intravenous injection between 2 to 6 hours prior to surgery. All subjects will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase A: LUM015 1.0 mg/kg: 5 participants received a single dose of LUM015 1.0 mg/kg administered by intravenous injection between 2 to 6 hours prior to surgery. All subjects will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase B: LUM015 1.0 mg/kg: 45 participants received a single dose of LUM015 1.0 mg/kg administered by intravenous injection between 2 to 6 hours prior to surgery. All subjects will have intraoperative imaging using the LUM 2.6 Imaging Device.
Period: Overall Study
Arm/Group | Phase A: No Dose | Phase A: LUM015 0.5 mg/kg | Phase A: LUM015 1.0 mg/kg | Phase B: LUM015 1.0 mg/kg
Started | 5 | 5 | 5 | 45
Completed | 5 | 5 | 5 | 44
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase A: No Dose: 5 participants were not administered with LLUM015 All participants will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase A: LUM015 0.5 mg/kg: 5 participants were administered with LLUM015 at 0.5 mg/kg by intravenous injection between 2 to 6 hours prior to surgery.
  All participants will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase A: LUM015 1.0 mg/kg: 5 participants were administered with LLUM015 at 1.0 mg/kg by intravenous injection between 2 to 6 hours prior to surgery.
  All participants will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase B: LUM015 1.0 mg/kg: 45 participants were administered with a single dose of LUM015 at 1.0mg/kg by intravenous injection between 2 and 6 hours prior to surgery. Patients will then undergo lumpectomy followed by LUM imagining of the lumpectomy cavity. Comprehensive shaves will be performed followed by LUM015 imagining of the resulting cavity and resection of LUM-imagining-positive cavity tissue.
- Total: Total of all reporting groups
Arm/Group | Phase A: No Dose | Phase A: LUM015 0.5 mg/kg | Phase A: LUM015 1.0 mg/kg | Phase B: LUM015 1.0 mg/kg | Total
Number analyzed (Participants) | 5 | 5 | 5 | 45 | 60
Age, Continuous [Median (Full Range); unit: years] | 69 [56 to 78] | 65 [48 to 70] | 59 [48 to 78] | 60 [44 to 79] | 60 [44 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 45 | 60
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 39 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 6 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 5 | 5
  White | 5 | 5 | 5 | 38 | 53
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 45 | 60
Cancer Histologic Type (from surgical excision) [Count of Participants; unit: Participants]
  Invasive Ductal Carcinoma with or without Ductal Carcinoma In Situ | 2 | 4 | 3 | 27 | 36
  Invasive Lobular Carcinoma with or without Ductal Carcinoma In Situ | 1 | 0 | 0 | 6 | 7
  Invasive Ductal Carcinoma and Invasive Lobular Carcinoma with or without Ductal Carcinoma In Situ | 0 | 0 | 1 | 1 | 2
  Pure Ductal Carcinoma In Situ | 2 | 1 | 1 | 9 | 13
  No Tumor Found | 0 | 0 | 0 | 2 | 2
Invasive Tumor Size in Largest Dimension [Median (Full Range); unit: cm] — Population: Not all patient tumors were measured.
  cm
    number analyzed (Participants) | 3 | 4 | 4 | 37 | 48
    (all) | 1 [0.6 to 1.3] | 1.85 [0.9 to 1.9] | 1.6 [0.4 to 2.5] | 1.2 [0.1 to 3.5] | 1.2 [0.1 to 3.5]
Patients with Node Positive Disease [Count of Participants; unit: Participants] — Population: Not all patients were diagnosed.
  Participants | 0 | 0 | 1 | 6 | 7
Tumor Receptors [Count of Participants; unit: Participants] — Population: Not all patients were diagnosed.
  Participants
    Her-2: number analyzed (Participants) | 4 | 4 | 4 | 30 | 42
    Her-2: Positives | 1 | 2 | 1 | 8 | 12
    Her-2: Negatives | 3 | 2 | 3 | 22 | 30
    Her-2: Neither triple negative nor triple positive | NA — Not applied | NA — Not applied | NA — Not applied | NA — Not applied | NA — Total not calculated because data are not available (NA) in one or more arms.
    Estrogen Receptor (ER): number analyzed (Participants) | 5 | 5 | 5 | 24 | 39
    Estrogen Receptor (ER): Positives | 5 | 5 | 4 | 19 | 33
    Estrogen Receptor (ER): Negatives | 0 | 0 | 1 | 5 | 6
    Estrogen Receptor (ER): Neither triple negative nor triple positive | NA — Not applied | NA — Not applied | NA — Not applied | NA — Not applied | NA — Total not calculated because data are not available (NA) in one or more arms.
    Progesterone Receptor (PR): number analyzed (Participants) | 5 | 5 | 5 | 24 | 39
    Progesterone Receptor (PR): Positives | 5 | 5 | 4 | 17 | 31
    Progesterone Receptor (PR): Negatives | 0 | 0 | 1 | 7 | 8
    Progesterone Receptor (PR): Neither triple negative nor triple positive | NA — Not applied | NA — Not applied | NA — Not applied | NA — Not applied | NA — Total not calculated because data are not available (NA) in one or more arms.
    All Triple Her-2, ER, PR: number analyzed (Participants) | 5 | 5 | 5 | 23 | 38
    All Triple Her-2, ER, PR: Positives | 1 | 2 | 1 | 0 | 4
    All Triple Her-2, ER, PR: Negatives | 0 | 0 | 1 | 4 | 5
    All Triple Her-2, ER, PR: Neither triple negative nor triple positive | 4 | 3 | 3 | 19 | 29
Menopausal Status [Count of Participants; unit: Participants]
  Post-menopause | 5 | 4 | 4 | 14 | 27
  Pre/Peri-menopause | 0 | 1 | 1 | 31 | 33
Mammographic Breast Density [Count of Participants; unit: Participants]
  Almost Entirely Fatty | 1 | 0 | 1 | 1 | 3
  Scattered Areas of Fibroglandular/Heterogeneously Dense | 2 | 1 | 0 | 18 | 21
  Heterogeneously Dense | 2 | 3 | 4 | 22 | 31
  Extremely Dense | 0 | 0 | 0 | 2 | 2
  Mixed Scattered Fibroglandular/Heterogeneously Dense | 0 | 1 | 0 | 2 | 3
Physical Examination Findings [Count of Participants; unit: Participants]
  Palpable Mass | 1 | 1 | 1 | 13 | 16
  No Palpable Mass | 4 | 4 | 4 | 32 | 44

OUTCOME MEASURES:

1. Primary Outcome: (Phase A Only) Selection of Dose of LUM015 to be Used in Future Breast Trials
Description: tumor-to-normal tissue signal ratio as a function of dose of LUM015
Time Frame: 1 day
Population: 5 patients not injected with LUM015, 5 patients injected with LUM015 at 0.5 mg/kg, and 5 patients injected with LUM015 at 1.0 mg/kg.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Phase A No LUM015: (Phase A only) 5 patients not injected with LUM015
- Phase A 0.5 mg/kg: (Phase A only) 5 patients injected with 0.5 mg/kg of LUM015
- Phase A 1.0 mg/kg: (Phase A only) 5 patients injected with 1.0 mg/kg of LUM015
Arm/Group | Phase A No LUM015 | Phase A 0.5 mg/kg | Phase A 1.0 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
Ratio | 2.1 (0.7) | 4.7 (2.0) | 4.2 (2.1)

2. Primary Outcome: (Phase B Only)Sensitivity and Specificity of the Lumicell Imaging System for Detecting Cancer
Description: Data from the participants in Phase A was used to develop an initial tumor detection algorithm that was then tested in Phase B. Thus, this endpoint is only applicable to the participants enrolled in the Phase B portion of the study.
  This endpoint measures the ability of the system to detect cancer as measured by sensitivity and specificity as defined below:
  Sensitivity = [number of true positives/(number of true positives + number of false negatives)] x 100% Specificity = [number of true negatives/(number of true negatives + number of false positives)] x 100%
  True positives = positive signal from imaging system and cancer found in tissue by pathology False positives = positive signal from imaging system and no cancer found in tissue by pathology True negatives = negative signal from imaging system and no cancer found in tissue by pathology False negatives = negative signal from imaging system and cancer found in tissue by pathology
Time Frame: 1 day
Population: Intent to treat population.
Measure: Mean (95% Confidence Interval); unit: percentage of measurements
Arm/Group | Phase B: LUM015 1.0 mg/kg
Number analyzed (Participants) | 45
percentage of measurements
  Sensitivity | 84 [79.5 to 88.5]
  Specificity | 73 [68.5 to 77.5]

3. Secondary Outcome: Number of Patients With Adverse Events as a Measure of Safety of the LUM Imaging System in Breast Cancer Subjects.
Description: Serious Adverse Events: Include adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
  Non-Serious Adverse Events: Adverse events that are not Serious Adverse Events.
Time Frame: Patients were evaluated for adverse events from time of injection until standard post-surgery follow-up visit. (Median 31 days after lumpectomy).
Population: Intent to treat population.
Measure: Count of Participants; unit: Participants
Groups:
- Phase B: LUM015 1. mg/kg: 45 participants were administered with a single dose of LUM015 at 1.0mg/kg by intravenous injection between 2 and 6 hours prior to surgery. Patients will then undergo lumpectomy followed by LUM imagining of the lumpectomy cavity. Comprehensive shaves will be performed followed by LUM015 imagining of the resulting cavity and resection of LUM-imagining-positive cavity tissue.
Arm/Group | Phase A: No Dose | Phase A: LUM015 0.5 mg/kg | Phase A: LUM015 1.0 mg/kg | Phase B: LUM015 1. mg/kg
Number analyzed (Participants) | 5 | 5 | 5 | 45
Participants
  Serious Adverse Event | 0 | 0 | 0 | 0
  Non-Serious Adverse Event | 0 | 0 | 0 | 5

ADVERSE EVENTS:
Time Frame: Patients were evaluated for adverse events from time of injection until standard psot-surgery follow-up visit. (Median 31 days after lumpectomy).
Groups:
- Phase A: No Dose: 5 participants were not administered with LUM015. All participants will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase A: LUM015 0.5 mg/kg: 5 participants were administered with a single dose of LUM015 at 0.5 mg/kg by intravenous injection between 2 and 6 hours prior to surgery. All participants will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase A: LUM015 1.0 mg/kg: 5 participants were administered with a single dose of LUM015 at 1.0 mg/kg by intravenous injection between 2 and 6 hours prior to surgery. All participants will have intraoperative imaging using the LUM 2.6 Imaging Device.
- Phase B: LUM015 1.0 mg/kg: 45 participants were administered with a single dose of LUM015 at 1.0 mg/kg by intravenous injection between 2 and 6 hours prior to surgery. Participants will then undergo lumpectomy followed by LUM imagining of the lumpectomy cavity. Comprehensive shaves will be performed followed by LUM015 imagining of the resulting cavity and resection of LUM-imagining-positive cavity tissue.
Arm/Group | Phase A: No Dose | Phase A: LUM015 0.5 mg/kg | Phase A: LUM015 1.0 mg/kg | Phase B: LUM015 1.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/45
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 5/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A: No Dose (N=5) | Phase A: LUM015 0.5 mg/kg (N=5) | Phase A: LUM015 1.0 mg/kg (N=5) | Phase B: LUM015 1.0 mg/kg (N=45)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post Procedural Hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Extravasation (General disorders) | 0 | 0 | 0 | 1
Suture Related Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
False positive readings may be associated with the LUM015 fluorescent signal extending beyond the tumor border, technical factors related to specimen processing and tissue sampling, and possible poor contact between the optical head and lumpectomy cavity wall, which may have reduced detection of fluorescent signal. This issues will be addressed in future clinical trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT02438358/Prot_SAP_000.pdf